CLINICAL TRIAL: NCT04330443
Title: Lung Ultrasound to Guide Surfactant Therapy
Acronym: ECOSURF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 136/2019
Record Dates: First submitted 2020-03-20; First posted 2020-04-01 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Experimental): The neonatologist-researcher (NR) performed the lung ultrasound at admission during the first hour of life. The neonatologist-assistant (NA) of the baby was not blinded to the result of the lung ultrasound. If the patient had a lung ultrasound score higher than >8 or when FiO2 exceeded 30% patient received surfactant therapy during in the first 72 hours of life
  Interventions: Procedure: Surfactant therapy
- Chest X Ray (No Intervention): The NR performed the LUS at admission/suspicion during the first hour of life. The NA was not blinded to the result of the LUS. Patient received surfactant therapy only when FiO2 exceeded 30% during the first 72 hours of life

INTERVENTIONS:
Procedure: Surfactant therapy — To study if lung ultrasound allows an earlier surfactant therapy (within the first 2 hours of life) compare to FiO2 and Chest X Ray
  Arms: Ultrasound group

SUMMARY:
Inclusion criteria are premature newborns under the gestational age (GA) of 32 weeks old with RDS, defined as the need of non invasive mechanical ventilation to keep peripheral oxygen saturation (SpO2) >90% and clinical signs of respiratory distress (polypnea, chest retractions, nasal flutter).

Exclusion criteria are non-acceptance of the informed consent, chromosomal abnormalities, complex congenital malformations, signs of congenital septic shock and mechanical ventilation or endotracheal surfactant prior to the lung ultrasound.

The main objective of the study is to determine if a diagnostic of respiratory distress syndrome guided by a lung ultrasound algorithm allow an earlier surfactant therapy (within the first 2 hours of life) comparing to chest X ray Secondary objectives were to assess FiO2 reached before surfactant therapy in patients surfacted according to the lung ultrasound score, the influence of the lung ultrasound algorithm regarding the respiratory evolution, and its differences comparing to the FiO2group. Respiratory evolution was defined as the need of mechanical ventilation, second dose of surfactant, duration of non invasive ventilation, number of days with oxygen requirements, length of stay in the neonatal intensive care unit, evolution to bronchopulmonary dysplasia and their progression to discharge from hospital.

Patients who met the inclusion criteria were randomly assigned to two groups. using the "random" function in MS-Excel XP® program. A total of 6 physicians enrolled participants, all them fully trained for the use of lung ultrasound. The principal investigator assigned participants to interventions, depending on the randomized list.

* Experimental Group 1: The neonatologist-researcher (NR) performed the lung ultrasond at admission during the first hour of life. The neonatologist-assistant (NA) of the baby was not blinded to the result of the lung ultrasound. If the patient had a lung ultrasound score higher than >8 or when FiO2 exceeded 30% patient received surfactant therapy during in the first 72 hours of life . This lung ultrasound threshold is the one with best diagnostic accuracy.
* Control Group 2: The NR performed the at admission/suspicion during the first hour of life. The NA was not blinded to the result of the ultrasound. Patient received surfactant therapy only when FiO2 exceeded 30% during the first 72 hours of life

DETAILED DESCRIPTION:
Inclusion criteria are premature newborns under the gestational age (GA) of 32 weeks old with RDS, defined as the need of non invasive mechanical ventilation to keep peripheral oxygen saturation (SpO2) >90% and clinical signs of respiratory distress (polypnea, chest retractions, nasal flutter).

Exclusion criteria are non-acceptance of the informed consent, chromosomal abnormalities, complex congenital malformations, signs of congenital septic shock and mechanical ventilation or endotracheal surfactant prior to the lung ultrasound.

The main objective of the study is to determine if a diagnostic of respiratory distress syndrome guided by a lung ultrasound algorithm allow an earlier surfactant therapy (within the first 2 hours of life) comparing to chest X ray Secondary objectives were to assess FiO2 reached before surfactant therapy in patients surfacted according to the lung ultrasound score, the influence of the lung ultrasound algorithm regarding the respiratory evolution, and its differences comparing to the FiO2group. Respiratory evolution was defined as the need of mechanical ventilation, second dose of surfactant, duration of non invasive ventilation, number of days with oxygen requirements, length of stay in the neonatal intensive care unit, evolution to bronchopulmonary dysplasia and their progression to discharge from hospital.

Patients who met the inclusion criteria were randomly assigned to two groups. using the "random" function in MS-Excel XP® program. A total of 6 physicians enrolled participants, all them fully trained for the use of lung ultrasound. The principal investigator assigned participants to interventions, depending on the randomized list.

* Experimental Group 1: The neonatologist-researcher (NR) performed the lung ultrasond at admission during the first hour of life. The neonatologist-assistant (NA) of the baby was not blinded to the result of the lung ultrasound. If the patient had a lung ultrasound score higher than >8 or when FiO2 exceeded 30% patient received surfactant therapy during in the first 72 hours of life . This lung ultrasound threshold is the one with best diagnostic accuracy.
* Control Group 2: The NR performed the at admission/suspicion during the first hour of life. The NA was not blinded to the result of the ultrasound. Patient received surfactant therapy only when FiO2 exceeded 30% during the first 72 hours of life

ELIGIBILITY:
Inclusion Criteria:

* premature newborns under the gestational age (GA) of 32 weeks old with respiratory distress syndrome

Exclusion Criteria:

* non-acceptance of the informed consent, chromosomal abnormalities, complex congenital malformations, signs of congenital septic shock and mechanical ventilation or endotracheal surfactant prior to the ultrasoundLUS

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Precocious surfactant administration | 2 monthts
  Number of patients which receive surfactant therapy during the first 2 hours of life

SECONDARY OUTCOMES:
assess FiO2 reached before surfactant therapy in patients surfacted according to the LUS score | 2 months
  assess FiO2 reached before surfactant therapy in patients surfacted according to the LUS score

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No